CLINICAL TRIAL: NCT03082573
Title: Open-label, Pilot Protocol of Patients With Rheumatoid Arthritis Who Were Treated With H.P. Acthar Gel After an Incomplete Response to Combinations of DMARDs and Biologic DMRADs
Brief Title: Efficacy, Radiographic and Laboratory Changes in Refractory Rheumatoid Arthritis Patients Treated With H.P. Acthar Gel
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iraj Sabahi Research Inc. (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IS2017
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Will be receiving the same background medications and H.P. Acthar gel 40 units twice weekly for 12 weeks.
  Patients in group A, can be cross over to group B on week 13 if disease is uncontrolled for continuation until week 24. If their disease is under control then they will continue with the same dosage until week 24.
  If the disease is under control, then tapering the steroid dosage can be attempted at the principal investigation's discretion.
  Interventions: Drug: H.P. Acthar gel
- Group B (Active Comparator): Will be receiving the same background medications and H.P. Acthar gel 80 units twice weekly for 12 weeks.
  if the disease is not under control, will continue with same dosage until week 24. If the disease is under control, will be given the option to reduce the dosage to 40 units twice weekly only if patient is suffering from H.P. Acthar gel related adverse effects.
  If the disease is under control, then tapering the steroid dosage can be attempted at the principal investigation's discretion.
  Interventions: Drug: H.P. Acthar gel

INTERVENTIONS:
Drug: H.P. Acthar gel — H.P. Acthar gel in treatment of Refractory RA
  Other Names: Repository Corticotropin Injection

SUMMARY:
This study will examine the clinical response, cytokine expression and joint imaging after addition of Acthar Gel. The hypothesis is that H.P. Acthar Gel is both safe and effective for treatment of patients with refractory rheumatoid arthritis (RA) and has different mechanism of action than steroids and other DMARDs.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a systemic inflammatory disease which causes premature mortality, disability and compromised quality of life in the industrialized and developing world. The prevalence of RA is believed to range from 0.5-1.0% in the general population. Over the past half century, many studies have found mortality to be increased in patients with established RA in comparison with the general population. Despite available treatment options for RA, some patients still have disease that is refractory to treatment and cannot achieve remission.

H.P. Acthar gel (adrenocorticotropic hormone gel) received FDA approval for treatment of a variety of diseases, including RA in 1952. The proposed efficacy of H.P. Acthar gel has been attributed to its ability to induce production of endogenous steroids and to bind melanocortin receptors on lymphocytes and other cells to modulate immunologic responses. The present study will examine the clinical response, cytokine production and joint imaging after addition of H.P. Acthar gel to confirm the efficacy, confirm different mechanism of action in comparison to steroids and other DMARDs by looking for post treatment changes in cytokine expression.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosis of RA with incomplete or failure to treatment described as either A or B A: Failure to achieve remission or low disease activity within 3 to 6 months of treatment with combination of methotrexate or other DMARDs therapy with a biologic DMARD in maximally tolerated doses within the usual therapeutic range.

   B- A requirement, in addition to DMARDs and biologic DMARDs, for chronic glucocorticoid therapy in a dose of greater than about 5 to 7.5 mg/day of prednisone or equivalent to achieve or maintain remission or low disease activity after 3 to 6 months of treatment.
2. Fluent in reading and writing in English language.
3. ≥ 21 years of age at the time of participation.

Exclusion Criteria:

1. Pregnancy
2. Presence if contraindications for treatment with H.P. Acthar gel including but not limited to any known history of scleroderma, osteoporosis, systemic fungal infections, ocular Herpes Simplex, recent administration of live or live attenuated vaccine (prior 6 months), recent surgery (prior 6 months), history of or the presence of a peptic ulcer, primary adrenocortical insufficiency, adrenal cortical hyperfunction; congestive heart failure (defined as New York Hear Association Functional Class I to IV, uncontrolled hypertension.
3. Previous use of ACTH preparations for treatment of nephrotic syndrome (including but not limited to H.P. Acthar gel and Synacthen®).
4. Previous history of sensitivity to ACTH preparations (including but not limited to H.P. Acthar gel and Synacthen®).
5. Previous history of sensitivity to porcine protein products.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
ACR 20 response ACR 20 response | Baseline to week 12
  Equal or greater than 20 % reduction in RA disease activity

SECONDARY OUTCOMES:
ACR 50 response | Baseline to week 24
  Equal or greater than 50 % reduction in RA disease activity
ACR 70 response | Baseline to week 24
  Equal or greater than 70 % reduction in RA disease activity
EULAR moderate response | Baseline to week 24
  Decline in the DAS 28 score by >1.2 (without reaching low disease activity) OR The decline of 0.6 to 1.2, plus reaching at least moderate disease activity (DAS28 <5.1).
EULAR good response | Baseline to week 24
  Decline in DAS 28 score must exceed 1.2 and result in the achievement of low disease activity (DAS28 <3.2).
Resolution of Powered Doppler Signal of MSKUS studies | Baseline to week 24
  Decline or resolution of synovitis detected in ultra sonographic examination of joints
Resolution of signs of active inflammation in MRI | Baseline to week 24
  Decline or resolution of synovitis, tenosynovitis or bone edema detected in MRI examination of joints
Reduction in Vectra DA Score | Baseline to week 24
  Decline in RA disease activity manifested as decline in Vectra DA Score
Correlation between MSKUS and MRI Imaging findings | Baseline to week 24
  Comparison between MSKUS and MRI imaging
Correlation between imaging findings and Vectra DA test | Baseline to week 24
  Comparison between MSKUS/MRI findings and Vectra DA test results

CONTACTS AND LOCATIONS:
Overall Officials: Iraj Sabahi, MD, Principal Investigator — Iraj Sabahi Research Inc.
Locations (2):
- United States (2):
  - Iraj Sabahi Research Inc, Pleasanton, California
  - Iraj Sabahi Research Inc, Turlock, California

IPD SHARING:
Plan to Share IPD: Undecided